CLINICAL TRIAL: NCT00529009
Title: Pharmacokinetic Investigation of UDCA in Bile and Serum
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Dr. Falk Pharma GmbH
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: URT-14/BIO
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Healthy
Keywords: PK analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: UDCA

SUMMARY:
To assess the bile acid composition of cystic bile and serum pharmaco¬kinetics after a 3-week treatment with UDCA and to correlate pharmacokinetic parameters of UDCA in bile and serum during steady state.

DETAILED DESCRIPTION:
see protocol

ELIGIBILITY:
Inclusion Criteria:

* PBC or healthy

Exclusion Criteria:

* pathology which does interfere with safety or PK of UDCA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Beuers, MD, Study Chair — University of Amsterdam
Locations (1):
- Beuers, Amsterdam, Netherlands

REFERENCES:
- [Result] Dilger K, Hohenester S, Winkler-Budenhofer U, Bastiaansen BA, Schaap FG, Rust C, Beuers U. Effect of ursodeoxycholic acid on bile acid profiles and intestinal detoxification machinery in primary biliary cirrhosis and health. J Hepatol. 2012 Jul;57(1):133-40. doi: 10.1016/j.jhep.2012.02.014. Epub 2012 Mar 10. PMID 22414767